CLINICAL TRIAL: NCT00454376
Title: Clinical and Psychometric Validation of a Disease-Specific Questionnaire Module in Assessing the Quality of Life of Patients With G.I.-Related Neuroendocrine Tumours
Brief Title: Disease-Specific Questionnaire in Assessing Quality of Life in Patients With Gastrointestinal-Related Neuroendocrine Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000537344; EORTC-QLQ-G.I.NET21; EU-20712; BNHFT-P4NET; EU-207101
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2008-11

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Lung Cancer; Metastatic Cancer; Neoplastic Syndrome
Keywords: metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; pulmonary carcinoid tumor; gastrinoma; insulinoma; WDHA syndrome; pancreatic polypeptide tumor; somatostatinoma; glucagonoma; liver metastases
MeSH Terms: conditions — Adenoma, Islet Cell; Lung Neoplasms; Neoplasm Metastasis; Neoplasms; Gastrinoma; Insulinoma; Vipoma; Somatostatinoma; Glucagonoma

INTERVENTIONS:
Other: questionnaire administration
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Questionnaires that measure quality of life may help doctors identify the effects of treatment and improve the ability to plan treatment for patients with gastrointestinal-related neuroendocrine tumors.

PURPOSE: This phase IV clinical trial is studying how well a disease-specific questionnaire works in assessing the quality of life of patients with gastrointestinal-related neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Test the scale structure, reliability, and validity of the gastrointestinal neuroendocrine tumor module (QLQ-G.I.NET21) in patients with gastrointestinal-related neuroendocrine tumors.

Secondary

* Determine the quality of life of patients using QLQ-C30 and the QLQ-G.I.NET21 before and after treatment.

OUTLINE: This is a multicenter study. Patients are stratified according to treatment (somatostatin analogue therapy or interferon therapy vs radionuclide therapy or chemotherapy vs ablative therapies [embolization or radiofrequency ablation] or liver resection).

Patients complete the EORTC C30 questionnaire, QLQ-G.I.NET21 module, and are evaluated for Karnofsky performance status at pretreatment, at 3 and 6 months after treatment, and then 2 weeks later. Patients also complete a clinical data and sociodemographic data form and debriefing questionnaire at pretreatment; a follow-up form at 3 months and 6 months after treatment; and a test-retest form 2 weeks later.

PROJECTED ACCRUAL: A total of 408 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroendocrine tumor OR characteristic radiological findings of neuroendocrine tumor with raised hormone levels in plasma or urine meeting any of the following criteria:

  * Primary disease in gut with liver metastases (with or without hormone secretion)
  * Primary disease in lung with liver or abdominal metastases (with or without hormone secretion)
  * Primary disease in pancreas with or without metastases (with or without hormone secretion)

PATIENT CHARACTERISTICS:

* Any Karnofsky performance status allowed
* Life expectancy ≥ 3 months
* Able to understand the questionnaire language
* Mentally fit to complete questionnaire
* No psychological, familial, sociological, or geographical condition that would limit study compliance
* No other concurrent malignancies except basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* More than 2 months since prior somatostatin analogue or interferon therapy (somatostatin therapy stratum)

  * Concurrent somatostatin analogue and/or interferon therapy allowed if dose stable over the past month
* More than 6 months since prior radionuclide therapy or systemic chemotherapy (radionuclide or systemic chemotherapy stratum)
* More than 6 months since prior ablative therapies (ablative therapy stratum)
* No concurrent participation in other quality of life studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Reliability, scaling, scale correlation, and clinical validity of the gastrointestinal neuroendocrine tumor module (QLQ-G.I.NET21)

SECONDARY OUTCOMES:
Response to change after various treatments

CONTACTS AND LOCATIONS:
Overall Officials: John K. Ramage, MD, Study Chair — Basingstoke and North Hampshire NHS Foundation Trust
Locations (16):
- Aarhus Universitetshospital - Aarhus Sygehus, Aarhus, Denmark
- Germany (2):
  - Charite - Campus Charite Mitte, Berlin
  - Klinikum der Universitaet Regensburg, Regensburg
- University Athens Alexandras Hospital, Athens, Greece
- Hadassah University Hospital, Jerusalem, Israel
- Clinical and Experimental Medicine at the University of Verona, Verona, Italy
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology - Warsaw, Warsaw, Poland
- Hospital Universitario San Carlos, Madrid, Spain
- Uppsala University Hospital, Uppsala, Sweden
- United Kingdom (6):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Aintree University Hospital, Liverpool, England
  - UCL Cancer Institute, London, England
  - King's College Hospital, London, England
  - Southampton General Hospital, Southampton, England
  - Royal Victoria Hospital, Belfast, Northern Ireland